CLINICAL TRIAL: NCT04450381
Title: Noninvasive Hemoglobin Testing in Prospective Blood Donors
Brief Title: Noninvasive Hemoglobin Testing, Prospective Blood Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SDBB0004
Record Dates: First submitted 2020-06-25; First posted 2020-06-29 (Actual); Results first posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Healthy; Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Test subjects (Experimental): All subjects are enrolled and receive Rad-67 Pulse oximeter & DCI Mini sensor for measurement of hemoglobin.
  Interventions: Device: Rad-67 Pulse oximeter & DCI Mini sensor

INTERVENTIONS:
Device: Rad-67 Pulse oximeter & DCI Mini sensor — Noninvasive pulse oximeter that measures hemoglobin

SUMMARY:
The objective of this clinical investigation is to evaluate the pulse oximeter devices for screening prospective blood donors. The purpose study is to report on the accuracy of noninvasive hemoglobin (SpHb) as compared to hemoglobin measurements obtained from a laboratory hematology analyzer in a blood donation setting.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Weight at least 110 pounds
* Subjects with the intention of being screened for eligibility to donate blood
* The subject has given written informed consent to participate in the study

Exclusion Criteria:

* Subjects with skin abnormalities at the planned application sites that may interfere with sensor application, per directions-for-use (DFU) or trans-illumination of the site, such as burns, scar tissue, infections, abnormalities, etc.
* Subjects unwilling and/or unable to remove nail polish or acrylic nails
* Subjects with blood cancers such as leukemia
* Subjects with hemoglobin disorders such as sickle-cell anemia and thalassemia
* Subjects with known history of infectious diseases such as HIV/AIDS, syphilis, hepatitis, etc.
* Subjects with self-disclosed/known pregnancy at the time of enrollment
* Subjects deemed not suitable for the study at the discretion of the investigator
* Excessive motion includes postural changes, making hand gestures, involuntary muscular movements, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Blood Bank - Site 1, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Subjects: All subjects are enrolled and receive the Pulse oximeter & sensor for measurement of hemoglobin.
  Rad-67 Pulse oximeter & DCI mini sensor: Noninvasive pulse oximeter that measures hemoglobin
Period: Overall Study
Arm/Group | Test Subjects
Started | 131
Completed | 125
Not Completed | 6
Not completed — Protocol Violation | 4
Not completed — Wrong device setting | 2

BASELINE CHARACTERISTICS:
Arm/Group | Test Subjects
Number analyzed (Participants) | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 106
  >=65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1
  Race: Asian | 16
  Race: Native Hawaiian or Other Pacific Islander | 2
  Race: Black or African American | 2
  Race: White | 76
  Race: More Than One Race | 6
  Race: Unknown or Not Reported | 3
  Race: Other: American | 1
  Race: Other: Assyrian | 1
  Race: Other: Mexican | 16
  Race: Other: Native American | 1
Region of Enrollment [Number; unit: participants]
  United States | 125

OUTCOME MEASURES:

1. Primary Outcome: Rad-67 Sensitivity
Description: Sensitivity of the the Rad-67 will be determined for its use in a blood donation center
Time Frame: Up to one hour per subject
Population: 2 subjects were excluded from analysis due to wrong device setting
Measure: Number; unit: percentage of sensitivity
Arm/Group | Test Subjects
Number analyzed (Participants) | 123
percentage of sensitivity | 44

2. Primary Outcome: Rad-67 Specificity
Description: Specificity of the the Rad-67 will be determined for its use in a blood donation center
Time Frame: Up to one hour per subject
Population: 2 subjects were excluded from analysis due to wrong device setting
Measure: Number; unit: percentage of specificity
Arm/Group | Test Subjects
Number analyzed (Participants) | 123
percentage of specificity | 86.73

ADVERSE EVENTS:
Time Frame: Up to one hour per subject
Arm/Group | Test Subjects
All-Cause Mortality (participants affected / at risk) | 0/131
Serious Adverse Events (participants affected / at risk) | 0/131
Other Adverse Events (participants affected / at risk) | 0/131

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT04450381/Prot_SAP_000.pdf